CLINICAL TRIAL: NCT04418037
Title: Digital Health Feedback System (DHFS) for Anti-Retroviral Therapy Medication Adherence and Transitions of Care Support During Hospital Admissions for Persons Living With HIV
Brief Title: DHFS for Medication Adherence Support During Hospital Admissions for Person Living With HIV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Gilead Sciences (Industry); ViiV Healthcare (Industry)
Responsible Party: Principal Investigator, Sara H. Browne, MD, MPH, Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 182100; R01MH110057 (NIH)
Record Dates: First submitted 2020-02-10; First posted 2020-06-05 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-11

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Single arm using the Digital Health Feedback System (Experimental): This protocol is designed to evaluate a novel technology that employs an ingestible sensor to detect medication ingestion for use by persons initiating or restarting antiretroviral (ARV) treatment for HIV infection during a hospital admission.
  Interventions: Device: Digital Health Feedback System(DHFS)

INTERVENTIONS:
Device: Digital Health Feedback System(DHFS) — We will investigate the feasibility of using the DHFS in hospitalized individuals living with HIV to support ARV adherence.

SUMMARY:
This study is a prospective single arm open label intervention study over 16 weeks using the DHFS and a telemedicine platform with persons living with HIV who are not virologically suppressed, admitted to UCSD Hillcrest Medical Center and initiating or restarting anti-retroviral therapy (ARVs). This proof of concept study will investigate the feasibility of using the DHFS in hospitalized individuals living with HIV to support ARV adherence. The Study intervention has an initiation phase of 2 weeks, a persistence phase of 14 weeks and a follow-up phase out to 48 weeks. Once study consent is obtained, the participant will receive a focused case navigation, psychiatric and substance abuse evaluation and will initiate digitized ARVs, either in hospital or at the AVRC within 14 days of hospital discharge, in collaboration with their providers. The study intervention will be considered to start from the point at which the DHFS is started. The study team will ensure the participants continue to utilize the DHFS both in hospital and after discharge. Following the 16 week intervention the study team will continue to follow participants to evaluate retention in care and viral suppression up to 48 weeks in collaboration with the outpatient care providers.

ELIGIBILITY:
Inclusion Criteria:

1. HIV seropositive status, as documented by positive licensed HIV antibody testing and a detectable viral load > 1000 copies/ml.
2. Persons admitted to UCSD Hillcrest Medical Center with an HIV associated diagnosis and to receive HIV care through UCSD Owen Clinic, FHCSD HIV Clinic or San Ysidro Health HIV Clinic post hospital discharge.
3. Persons initiating or continuing treatment for HIV infection by their HIV provider, that includes either:

   1. Dolutegravir/Tenofovir alafenamide/Emtricitabine: IS-DTG/TAF/FTC (Tivicay® and Descovy®)
   2. Bictegravir/ Tenofovir alafenamide/Emtricitabine: IS-BIC /TAF/FTC (Biktarvy®)
   3. Darunavir/Cobistat/Emtricitabine/Tenofovir alafenamide: IS-DRV/C/F/TAF (Symtuza™)
4. Eligible for antiretroviral medications and in possession of prescriptions for above noted study eligible regimens.
5. Laboratory values obtained by screening laboratories within 30 days of entry:

   1. Absolute neutrophil count (ANC) ≥ 1,000/mm3.
   2. Hemoglobin ≥ 7.0 g/dL.
   3. Platelet count ≥ 50,000/mm3.
   4. AST (SGOT), ALT (SGPT), and alkaline phosphatase ≤ 5 x ULN.
   5. Total bilirubin ≤ 3 x ULN and direct bilirubin.
   6. Estimated GFR by Cockcroft-Gault equation of greater than 30 ml/min.
6. Females of childbearing potential (defined as girls who have reached menarche or women who have not been post-menopausal for at least 24 consecutive months, i.e. who have had menses within the preceding 24 months, or have not undergone surgical sterilization (e.g. hysterectomy, bilateral oophorectomy, or salpingotomy) must have a negative serum or urine pregnancy test performed within 72 hours prior to study entry.

   If participating in activity that could lead to pregnancy, the participant must use at least one of the following forms of contraception throughout the protocol and for 6 weeks after stopping the IS-ARV medications.
   * Condoms (male or female) with a spermicidal agent
   * Diaphragm or cervical cap with spermicide
   * IUD
   * Oral contraception. Condoms in addition to other methods are highly recommended because their appropriate use is the only contraception method effective for preventing HIV-1 transmission.
7. Men and women age ≥ 18 years.
8. Basic competency in understanding written and verbal information as it applies to DHFS use. English and Spanish will be used for study documents and communication.
9. Ability and willingness to follow all protocol requirements.
10. Ability to use mobile device per investigator determination, and to wear PDH wearable sensor (i.e., no skin conditions precluding use).
11. Ability and willingness of participant to give written informed consent.

Exclusion Criteria:

1. Female who is pregnant, breast-feeding, or of childbearing potential and disagrees to use contraception throughout the study period.
2. Use of any of the prohibited medications or other non-informed medications (Section 5.5.2) within 30 days of study entry (Day 0).
3. Known allergy/sensitivity to any of the study drugs.
4. Known sensitivity to skin adhesives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
An accurate measure of medication taking adherence captured by the DHFS | 16 weeks
  The number of doses ingested as captured by the DHFS over the number of doses prescribed, adjusted for positive detection accuracy (PDA). The system positive detection accuracy (PDA), based on prior studies, will allow an accurate measure of adherence with CI calculated.

SECONDARY OUTCOMES:
Achieving <90% adherence as detected by DHFS over the study intervention (weeks 0-16). | 16 weeks
  Participants with <90% adherence as detected by DHFS over the study intervention will be identified.
Percentage of participants who require adherence support to maintain adherence over 90% during weeks 0-16. | 16 weeks
  Percentage of participants who require adherence support to maintain adherence over 90% will be calculated.
Satisfaction rating for DHFS use for HIV treatment as 'satisfactory' or higher. | 16 weeks
  Characterize participant responses to study questionnaires on usability and exit questionnaire and summarize information regarding patient experience with the DHFS.

CONTACTS AND LOCATIONS:
Overall Officials: Sara H Browne, MD MPH, Principal Investigator — UC San Diego
Locations (1):
- UCSD AntiViral Research Center, San Diego, California, United States

DOCUMENTS (1):
  • Informed Consent Form (2022-02-08): https://cdn.clinicaltrials.gov/large-docs/37/NCT04418037/ICF_000.pdf